CLINICAL TRIAL: NCT07010679
Title: Development and Pilot Testing of a Patient-Centered Clinical Decision Support for Chronic Rhinosinusitis
Brief Title: Treatment Decision-Making Among Patients With Chronic Rhinosinusitis
Acronym: CRS-AID
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Shinyi Wu, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UP-22-00453-AM008; APP-25-00437 (Other: University of Southern California IRB)
Record Dates: First submitted 2025-05-15; First posted 2025-06-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Rhinosinusitis (CRS)
Keywords: Patient decision aid; Patient-centered Clinical Decision Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will use the patient centered clinical decision support (PC CDS) tool in addition to receiving standard care.
  Interventions: Other: Patient Centered CRS Treatment Decision Support
- Control Group (No Intervention): Participants in this group will receive standard care, which includes informational handouts about CRS management.

INTERVENTIONS:
Other: Patient Centered CRS Treatment Decision Support — The intervention is a web-based tool that includes:
  * Educational content and Frequently Asked Questions (FAQ) about CRS and treatment options
  * Patient stories from CRS patient interviews with artificial intelligence-assisted narrative writing
  * A communication tool to support discussions between patients and their doctors
  * Culturally tailored components, including Chinese language options and culturally relevant narratives Participants will be introduced to the PC CDS during a routine clinic visit or through a scheduled virtual meeting. They will use the tool before making treatment decisions. The tool is designed to be user-friendly and accessible across devices.
  Arms: Intervention Group

SUMMARY:
This project aims to develop and pilot-test a bilingual, patient-centered clinical decision support (PC CDS) web application for individuals with chronic rhinosinusitis (CRS), a condition affecting 16% of U.S. adults annually and significantly impacting quality of life. While endoscopic sinus surgery (ESS) is a recommended treatment for medically refractory cases, many patients experience barriers that lead to surgical hesitancy. Prior research at USC revealed significant disparities in ESS uptake (Odds Ratio = 7.92; 95% Confidence Interval: 2.95-21.28), highlighting the need for more tailored decision support.

The PC CDS will include educational resources, Large Language Model-assisted patient narratives, and a provider communication module to facilitate shared decision-making (SDM). The study has three aims: (1) to develop the tool; (2) to evaluate its feasibility in a randomized controlled trial with 50-60 patients from USC clinics; and (3) to assess outcomes using surveys and interviews. Participants will be randomized into either a control group (receiving standard CRS informational handouts) or an intervention group (receiving standard care plus the PC CDS tool).

Quantitative surveys will measure treatment choice, decision quality, SDM involvement, CRS knowledge, provider trust, and care satisfaction. Qualitative interviews will explore participants' healthcare journeys and experiences with the tool. Guided by experts in health technology and rhinology and in collaboration with a Patient Advisory Group, the study aims to ensure patient-centered design and lay the groundwork for future implementation and external funding (e.g., AHRQ).

DETAILED DESCRIPTION:
This research aims to develop and pilot-test a patient-centered clinical decision support (PC CDS) web application specifically for patients with chronic rhinosinusitis (CRS). CRS, which affects approximately 16% of U.S. adults annually, significantly impacts quality of life (QOL). Endoscopic sinus surgery (ESS) is a recommended treatment for those unresponsive to medical therapy; however, many patients face unique barriers that contribute to surgical hesitancy and suboptimal outcomes. A previous study conducted at the University of Southern California (USC) revealed significant differences in the likelihood of undergoing ESS among patient subgroups (Odds Ratio = 7.92; 95% Confidence Interverval: 2.95-21.28; p < 0.001). To address these disparities, the proposed PC CDS will integrate patient-centered support components tailored for individuals hesitant or resistant to ESS, including educational resources, Large Language Model-assisted patient narratives, and a patient-provider communication feature within a bilingual decision aid.

The project includes three primary aims: (1) develop the PC CDS to facilitate shared decision-making (SDM) between patients and clinicians, with the goal of reducing surgical hesitancy and improving outcomes; (2) recruit 50-60 medically refractory CRS patients from USC clinics in Los Angeles for a randomized controlled feasibility trial comparing standard care to the PC CDS intervention; and (3) assess patient healthcare journey outcomes, as well as the acceptability and usability of the PC CDS, through pre- and post-intervention evaluations using both quantitative and qualitative methods.

Participants will be randomly assigned to one of two groups:

Control Group: Will receive standard care, including informational handouts on CRS management.

Intervention Group: Will receive access to the PC CDS tool in addition to standard care.

Data will be collected through surveys and interviews to evaluate healthcare experiences and the influence of the PC CDS tool.

Surveys (Quantitative Measures):

To evaluate whether the PC CDS affects treatment decision-making in CRS care, participants in both groups will complete surveys capturing:

Treatment selection (surgery or no surgery) Quality of decision-making experience, including alignment with patient goals Level of involvement in shared decision-making Knowledge of CRS and trust in the healthcare provider Overall satisfaction with care

Interviews (Qualitative Measures):

Trained interviewers will conduct qualitative interviews with all participants to gain deeper insight into healthcare experiences, engagement with the educational materials or PC CDS tool, and factors influencing treatment decisions.

The research team, led by experts in health technology and rhinology, will collaborate with a Patient Advisory Group to ensure the tool is patient-centered and responsive to community needs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patient receiving care at a USC otolaryngology clinic located in Los Angeles, Glendale, La Cañada, or Arcadia
* Diagnosis of chronic rhinosinusitis (CRS) as defined by the American Academy of Otolaryngology-Head and Neck Surgery criteria
* Medically refractory CRS (i.e., persistent symptoms despite appropriate medical therapy)
* Considered a candidate for endoscopic sinus surgery (ESS) by the treating otolaryngologist
* English- or Chinese-speaking
* Able and willing to provide informed consent
* Access to a smartphone, tablet, or computer with internet connection

Exclusion Criteria:

• Not offered endoscopic sinus surgery (ESS) as a treatment option by the treating otolaryngologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Choosing Endoscopic Sinus Surgery (ESS) vs. Nonsurgical Management at 4-Month Follow-up | Up to 4 months post-enrollment
  The primary outcome will be the proportion of participants in each study arm (PC CDS intervention vs. standard care control) who elect to pursue either endoscopic sinus surgery (ESS) or nonsurgical treatment within four months following enrollment. Treatment decisions will be assessed via self-report and confirmed through medical record review. Data will be summarized as percentages for each group, and between-group differences will be compared using chi-square or Fisher's exact tests. This measure will evaluate the effect of the PC CDS tool on surgical acceptance rates among patients with medically refractory chronic rhinosinusitis (CRS).
Decision Concordance as Measured by an Adapted Decision Quality Instrument for Chronic Rhinosinusitis (DQI-CRS) | At 4 weeks post-enrollment
  Decision concordance will be assessed using an adapted version of the Decision Quality Instrument (DQI) tailored to chronic rhinosinusitis (CRS). Participants will identify their top treatment goals and report the treatment option they ultimately selected (e.g., surgery or continued medical management). Concordance will be evaluated by comparing the stated treatment preference (based on ranked goals) to the actual treatment decision. A concordance score will be calculated as the percentage of participants whose treatment choice matches their top-ranked goals and concerns. Higher scores reflect better alignment between patients' preferences and treatment decisions. The adapted concordance assessment will be reviewed by clinical experts and a Patient Advisory Group prior to administration.
Shared Decision-Making Experience as Measured by the 9-item Shared Decision Making Questionnaire (SDM-Q-9) | At 4 weeks post-enrollment
  Shared decision-making experience will be assessed using the 9-item Shared Decision Making Questionnaire (SDM-Q-9), a validated patient-reported measure that evaluates the extent to which patients perceive involvement in the clinical decision-making process. Each item is rated on a 6-point Likert scale ranging from 0 (completely disagree) to 5 (completely agree), yielding a total score between 0 and 45. Scores will be linearly transformed to a 0-100 scale, with higher scores indicating a more positive SDM experience. The SDM-Q-9 will be administered 4 weeks after enrollment to evaluate the impact of the PC CDS tool on patient-perceived engagement in decision-making for CRS treatment.
CRS Knowledge Score Based on a 10-Item Investigator-Developed Questionnaire | At baseline and at 4 weeks post-enrollment
  Patient knowledge of chronic rhinosinusitis (CRS) will be assessed using a 10-item questionnaire developed by the investigative team. The questionnaire includes multiple-choice and multi-response items covering key domains of CRS knowledge, such as disease definition, diagnostic criteria, treatment options (including endoscopic sinus surgery), associated risk factors, and expected surgical outcomes. One question uses a multi-select format in which the correct answer requires selecting all appropriate responses. Each item is scored as correct or incorrect, with one point awarded for each correct answer (including full accuracy on the multi-select item), resulting in a total score ranging from 0 to 10. Higher scores indicate greater factual knowledge about CRS and its treatment.
Trust in Physician as Measured by the 10-item Wake Forest Physician Trust Scale (WFPTS) | At baseline and at 4 weeks post-enrollment
  Trust in the treating physician will be assessed using the 10-item Wake Forest Physician Trust Scale (WFPTS), a validated patient-reported measure that evaluates interpersonal trust across multiple domains, including fidelity, competence, honesty, confidentiality, and dependability. Each item is rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), with total scores ranging from 10 to 50. Higher scores indicate greater trust in the physician. The WFPTS has demonstrated strong psychometric properties, including high internal consistency (Cronbach's alpha = 0.93) and unidimensional factor structure, as evidenced by exploratory and confirmatory factor analyses. The scale has been adapted and validated in various cultural contexts, supporting its applicability across diverse patient populations.

SECONDARY OUTCOMES:
Disease-specific quality of life related to chronic rhinosinusitis (CRS) as measured by the SinoNasal Outcome Test - 22 items | at baseline and also either 1 and 3 months after surgery, or 2 and 4 months after baseline if patient do not undergo surgery
  Disease-specific quality of life related to chronic rhinosinusitis (CRS) will be assessed using the Sino-Nasal Outcome Test-22 (SNOT-22), a validated 22-item patient-reported outcome measure. Each item is scored on a 6-point Likert scale ranging from 0 ("No problem") to 5 ("Problem as bad as it can be"), resulting in a total score range of 0 to 110. Higher scores indicate worse sinonasal-related quality of life. The SNOT-22 includes domains such as nasal symptoms, sleep function, and emotional impact. For participants who undergo surgery, the instrument will be administered at 1 and 3 months following the surgical date. For participants who do not undergo surgery, the SNOT-22 will be administered at 2 and 4 months following study enrollment to provide comparable longitudinal assessment. This outcome will be used to evaluate clinical effectiveness of the PC CDS tool in supporting informed treatment decisions and improving CRS-related outcomes.
Patient-Reported Satisfaction with CRS Knowledge and Treatment Decision Confidence | At 4 weeks post-enrollment
  Patient satisfaction with knowledge and information received regarding chronic rhinosinusitis (CRS), as well as treatment preferences and confidence in decision-making, will be assessed using a custom, investigator-developed questionnaire. The instrument consists of six items addressing the following areas: (1) satisfaction with current knowledge about CRS and treatment options; (2) satisfaction with information received to date; (3) self-reported need for additional information; (4) treatment options currently being considered (lifestyle modifications, medical management, surgery); (5) confidence in treatment decision; and (6) awareness of CRS subtype (e.g., CRS with or without nasal polyps). Responses are collected using categorical and Likert-style options. Descriptive analyses will be used to summarize patient-reported levels of satisfaction, information needs, decision confidence, and treatment readiness.

CONTACTS AND LOCATIONS:
Overall Officials: Shinyi Wu, PhD, Principal Investigator — University of Southern California
Locations (1):
- Keck Medicine of USC, Arcadia, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying published results, including demographics, outcomes, and survey responses, will be made available to qualified researchers following publication of primary study findings.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be shared beginning 6 months after publication of the main results and will be available for up to 36 months thereafter.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal and agree to a data use agreement. Requests should be submitted to the study principal investigator via institutional email.